CLINICAL TRIAL: NCT05438290
Title: A Phase I, Open Label Study Employing the Topical Immunomodulator Diphencyprone to Treat Cutaneous Neurofibromas Associated With NF1
Brief Title: DPCP to Treat Cutaneous Neurofibromas Associated With NF1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nicholas Gulati (Other)
Responsible Party: Sponsor-Investigator, Nicholas Gulati, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-00650
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Cutaneous Neurofibroma
Keywords: NF1; neurofibromatosis type 1; neurofibromatosis; NF
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses | interventions — diphenylcyclopropenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DPCP (Experimental): 0.4% ointment
  Interventions: Drug: DPCP

INTERVENTIONS:
Drug: DPCP — topical immunomodulator
  Other Names: diphencyprone

SUMMARY:
Neurofibromatosis type 1 (NF1) is the most common genetic tumor predisposition syndrome, affecting up to 1 in 2500 individuals. Cutaneous neurofibromas are benign with self-limited growth; however, tumor burden may be excessive, tumors do not regress, and they can be disfiguring, painful, and itchy. Currently, the only treatment is surgery or laser ablation; however, outcomes are limited by the number of tumors that can be simultaneously removed, operating room availability, and painful recovery, with significant risk of regrowth. There is a strong need for noninvasive topical treatments for cutaneous neurofibromas. Diphencyprone (DPCP) is a "hapten" medication, a small molecule that activates the immune system when applied topically, which has been investigated as a cutaneous immunotherapy for other skin conditions.

This is an open label Phase I study looking at safety and tolerability of this treatment as a primary endpoint, and tumor treatment as a secondary endpoint. Approximately 30 subjects will be enrolled at a single center within the US. Subjects with a clinical diagnosis of NF1 who have measurable disease and at least 4 cutaneous neurofibromas, will have DPCP applied topically to their neurofibromas once weekly for 10 weeks.

DETAILED DESCRIPTION:
Each subject after consent will undergo a biopsy of one cutaneous neurofibroma prior to treatment. The participant will then undergo a sensitization treatment to "normal" skin as well as one neurofibroma to activate the immune system against the trial drug. 14 days after sensitization, patients will begin the first of 10 weekly treatment doses to a minimum of 3, up to 20 cutaneous neurofibromas. The participant may require up to 2 additional sensitization exposures. When the investigator has determined that sensitization has occurred, each subject will have a skin biopsy of one treated neurofibroma 3 days after initial treatment on Day 17 in order to investigate cellular and molecular effects of the treatment. The remainder of treatments will be applied once weekly on days 21, 28, 35, 42, 49, 56, 63, 70, and 77. The followup visit will occur on Day 107. Tumors will be photographed at screening and at each treatment visit, and in addition, whole body photography will be performed on Day 0 and Day 107 to assess for off-target effects on cutaneous neurofibromas that were not directly treated. On Day 107, a third cutaneous neurofibroma will be biopsied for molecular and immunohistopathological outcomes.

ELIGIBILITY:
Inclusion Criteria

* Clinically diagnosed NF1 as per the expertise of the study team.
* At least four cutaneous neurofibromas greater than 4 mm in size that are able to be biopsied.
* Age ≥ 18 years.
* Ability to understand and the willingness to sign a written informed consent.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  1. Has not undergone a hysterectomy or bilateral oophorectomy; or
  2. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria

* Subjects may not be receiving any other investigational agents.
* Subjects taking any of the following systemic therapies within 2 weeks of enrollment: corticosteroids, immunosuppressants, and/or any other medications (systemic or topical) that may affect the outcome of the study in the opinion of the investigator.
* Subjects with any underlying diseases or dermatological conditions of the affected areas that require the use of interfering topical or systemic therapy, or that may impair immune responses such as HIV or lymphadenectomy of the axillary lymph node basin that drains the skin where DPCP is to be applied.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DPCP, or any of the other components of the DPCP ointment formulation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a grade 3 adverse event | at Day 77 or 107
  Safety of DPCP will be measured as the proportion of subjects with a grade 3 on the Common Terminology Criteria for Adverse Events (CTCAE) criteria. Specifically, the safety of DPCP will be assessed as per CTCAE for eczema, version 5.0.
Symptom standardized assessment scale | at Day 77 or 107
  Tolerability of DPCP will be measured by the subjective response of patients who experience symptoms directly related to the therapy. Specifically, the subject will report their own symptoms of local tolerability based on a standardized assessment scale. The subject will assess pain, stinging, burning, and pruritus using a 4-point scale (0 none, 1 mild, 2 moderate, 3 severe) for each treated target lesion. Each of the four domains will be graded on the 4-point scale, each domain range from 0-16, with higher score indicating more severe symptoms. There is no overall score.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Gulati, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Rebecca Brown, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Specify Other Mechanism PI to be contacted
URL: https://www.mountsinai.org/care/neurology/services/neurofibromatosis

DOCUMENTS (1):
  • Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT05438290/ICF_000.pdf